CLINICAL TRIAL: NCT02338063
Title: Eliciting Affect in Teens in a Virtual World (Project AVATAR)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0079-10; 5R42MH087322-03 (NIH)
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: HIV Infections
Keywords: Adolescent Risk Behavior; Emotion Regulation; Health Promotion; Intervention; Mental Health
MeSH Terms: conditions — HIV Infections; Emotional Regulation; Psychological Well-Being | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Virtual Reality
  Interventions: Behavioral: Virtual Reality
- 2 (Experimental): Health Promotion
  Interventions: Behavioral: Health Promotion

INTERVENTIONS:
Behavioral: Virtual Reality — 4-session group intervention including affect management training as well as sexual health skills training to prevent the transmission of HIV. Group will practice skills using 3-D goggles for some activities.
  Other Names: IVRE intervention
  Arms: 1
Behavioral: Health Promotion — 4-session group intervention including affect management training as well as sexual health skills training to prevent the transmission of HIV. Group will practice skills using traditional role-plays for some activities.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether immersive virtual reality technology is an effective intervention tool for HIV Prevention with adolescents.

DETAILED DESCRIPTION:
The project will examine the use of immersive virtual reality technology as an intervention tool for HIV Prevention with adolescents. Adolescents are at risk for contracting HIV while affect dysregulation is common among adolescents. Research has demonstrated connections between poor affect management abilities and risky sexual behavior among adolescents. This research suggests that the ability to regulate one's emotions is key to avoiding risk behaviors and that adolescents are at greater risk for poor affect management skills. Fortunately, these skills can be taught via teaching and modeling, making them an excellent target for intervention, which has previously been approached through role-playing. Immersive virtual reality offers many advantages over group based role-plays, used in HIV prevention interventions for adolescents, in its ability to simulate real-world environments and enhance the impact of HIV prevention interventions. Immersive virtual reality is a promising technology for giving teens the opportunity to experientially practice using effective affect regulation skills in a highly realistic, context specific virtual environment. Additional benefits of this technology will likely be increased engagement and retention in HIV prevention interventions among young adolescents. The overall aims of Phase I and Phase II of this project are to develop, refine, and evaluate virtual reality environments for adolescents targeting affect management. In Phase I, the research team developed and refined an immersive virtual environment that elicited affect in a high-risk situation. The final immersive virtual reality environments (completed in Phase II) can be used by health promotion interventionists in conjunction with an HIV prevention intervention manual as a means to elicit affect and provide adolescents with a "real world" environment in which to practice emotion regulation skills related to substance use and HIV prevention. These aims will be achieved through the collaboration of researchers at Rhode Island Hospital/Brown and Virtually Better, Inc. a small business that specializes in creating immersive virtual reality environments for treatment, education, and training purposes. This tool will represent a significant advance in the way in which affect regulation skills are practiced and honed, currently achieved via role plays or imaginal exposure, by increasing the salience of cues used to elicit affect, thus making it highly marketable to interventionists, schools, and mental health clinicians.

ELIGIBILITY:
Inclusion Criteria:

- 7th & 8th graders at participating public schools.

Exclusion Criteria:

* Adolescent is illiterate.
* Adolescent has parent/guardian who does not speak English.
* Adolescents has high risk of motion sickness.
* For Phase II only, previous participation in Project Trac or Phase I.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2010-05; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Adolescent-reported self-efficacy for HIV prevention behaviors | 3 months

SECONDARY OUTCOMES:
Adolescent-reported condom use self-efficacy | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States